CLINICAL TRIAL: NCT00221910
Title: Does Ultrasound Guidance Improve the Success of Sciatic Nerve Block at the Popliteal Fossa? A Prospective, Randomized, Controlled Trial.
Brief Title: Use of Ultrasound in Lower Extremity Blocks.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UHN02-0771-B
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2005-03

CONDITIONS: Regional Anesthesia
MeSH Terms: interventions — High-Energy Shock Waves

INTERVENTIONS:
Procedure: Ultrasound

SUMMARY:
Nerve "freezing" injections of the leg are very useful in providing anesthesia and pain relief for knee and ankle surgery. However, current nerve "freezing" techniques are "blind". As a result, they are not always successful and may cause complications, albeit infrequent.

The objective of the current study is to determine any advantage in performing these "freezing" injections under direct ultrasound guidance, to "visualize" the nerves. We feel that by developing this technique, it will allow us to perform these procedures with greater success and fewer complications.

DETAILED DESCRIPTION:
This study is a randomised controlled trial. Its objective is to compare results and complications between two techniques of nerve localisation for nerve blocks of the lower limb. We have developed a real-time, image guided approach to nerve blocks of the lower extremities in three locations: the femoral nerve in the groin and the sciatic nerve in the buttock and/or popliteal fossa. We have used ultrasound imaging to locate and asess the nerves of the lower extremities and to use it as a real-time guidance for performance of lower extremity blocks in patients undergoing orthopaedic procedures. The results of our previous study will be presented as a case series reporting anatomical appearance of the nerves studied, time for block performance and success rates. In this study we aim to compare these parambeters between standard and ultrasound techniques of lower extremity block, to show any advantage.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* ASA physical status I-III
* 18-85 years of age, inclusive
* 50-110 kg, inclusive
* 150 cm of height or grater
* Scheduled for elective foot or ankle surgery

Exclusion Criteria:

* Contraindications to sciatic nerve block (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the popliteal area)
* Significant peripheral neuropathy or neurologic disorder affecting the lower extremity
* Pregnancy
* Contraindications to, allergies to, and/or past adverse reactions to local anesthetics
* History of alcohol or drug dependency/abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada